CLINICAL TRIAL: NCT05668442
Title: Online Physical Exercise and Group Sessions to Increase and Maintain Physical Activity in Individuals With Type 2 Diabetes: A Single-Arm Feasibility Study
Brief Title: Feasibility of an Online Exercise Community Among Individuals With Type 2 Diabetes
Status: Completed | Type: Observational
Sponsor: Mathias Ried-Larsen (Other)
Responsible Party: Sponsor-Investigator, Mathias Ried-Larsen, Principal Investigator, Rigshospitalet, Denmark
Organization: Rigshospitalet, Denmark (Other)
Other Study IDs: H-21062951
Record Dates: First submitted 2022-11-18; First posted 2022-12-29 (Actual); Last update posted 2023-01-03 (Actual); Status verified 2022-12

CONDITIONS: Type 2 Diabetes; Type2diabetes; Diabetes Mellitus, Type 2; Type2 Diabetes Mellitus
Keywords: Obesity; Feasibility; Physical activity; Type 2 diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Obesity; Motor Activity

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Behavioral: Online exercise and group meetings — The intervention consists of 8 weeks of 30 minutes of online supervised high intensity physical exercise followed by 30 minutes of online group meeting once a week in Microsoft Teams. The program consist of a short warm-up, followed by interval.-based physical activity including bodyweight aerobic and strength training, followed by stretching.
  Following the online exercise session, participants will be sent out in smaller break-out rooms in Microsoft Teams. The online group meeting sessions are intended to serve as a platform for group discussion evaluation of weekly physical acitvity.
  Each online group will be facilitated by a participant. All participants will be encouraged to set physical activity goals to increase habitual physical activity As a part of the intervention, participants will wear a Garmin Vivofit 4 activity watch or a Garmin 245 watch.

SUMMARY:
The aim of this study is to evaluate the feasibility, fidelity and acceptability of an 8-week high intensity online physical exercise combined with online group meetings and supported with an activity tracker in individuals with type 2 diabetes. The design of the intervention will be developed using a co-creation approach. The intervention consist of eight weeks of 30 minutes online physical exercise followed by 30 minutes of online group meeting in Microsoft Teams once a week. Outcomes includes pre-defined research progression criteria and secondary outcomes of physical and mental health and participant feedback.

DETAILED DESCRIPTION:
The study is designed as a one-armed feasibility for the reason that the progression criteria are linked to the intervention. No blinding will be applied in the study.

The study will be carried on the Centre for Physical Activity Research, Rigshospitalet, Denmark. Reporting of the study will be following the CONSORT extension to a randomized pilot and feasibility trials.

Participants will be recruited from the Capital Region of Denmark and Region Zealand using different recruitment strategies followed by a telephone screening with the project coordinator.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with type 2 diabetes
* Access to a device such as a computer, tablet, or a smart phone

Exclusion Criteria:

* Contraindications to exercise, for example heart conditions, complications/injuries in the locomotive apparatus
* Advised to not exercise by medical doctor
* Current participation in other intervention trials

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: All participants were recruited within the Capital of Region of Denmark and Region of Southern Zealand. Males and females >18 years old and diagnosed with T2D were included. Furthermore, the participants were required to have access to a device such as a computer, tablet, or a smart phone. The exclusion criteria were contraindications to exercise (e.g., unstable cardiovascular disease, complications/injuries in the locomotive apparatus). Furthermore, participants were excluded if they were advised not to exercise by a doctor or already participating in other intervention trials.
Sampling Method: Non-Probability Sample
Enrollment: 24 (Actual)
Dates: Start 2020-11-21 (Actual); Primary Completion 2022-06-06 (Actual); Study Completion 2022-06-06 (Actual)

PRIMARY OUTCOMES:
Research Progression Criteria | 8 weeks
  Research Progression Criteria obtained through self-reported data from weekly questionnaires organized into the following categories:
  Participant recruitment Completion of intervention Adherence to online physical exercise Adherence to the group meeting Adherence to goal setting Difficulty in participating in the objectively measured physical activity Improvement of physical activity Adverse events
Participant Recruitment | 3 months
  Evaluation of participant recruitment was made by calculating number of participants recruited within three months.
Completion of intervention | 10 weeks
  Evaluation of completion of the intervention was made by calculating the percentage of participants who provided baseline and postintervention data out of the total number of participants at baseline
Adherence to online physical exercise | 8 weeks
  Evaluation of adherence to online physical exercise, participants received weekly web-based questionnaires instantly after the online physical exercise to respond whether they attended the session.
  Adherence to online physical exercise was calculated by counting the number of completed online meetings separately, divided by the eight planned sessions.
Adherence to online meeting | 8 weeks
  Evaluation of adherence to online group meetings, participants received weekly web-based questionnaires instantly after the online meeting to respond whether they attended the session.
  Adherence to online meeting was calculated by counting the number of completed online meetings separately, divided by the eight planned sessions.
Adherence to goal setting | 8 weeks
  During the 8-week intervention, participants wrote down a weekly activity goal for the forthcoming week and if they completed the activity goal from the previous week.
Difficulty in participating in the objectively measured physical activity | 8 weeks
  Difficulty in participating in the objectively measured physical activity was evaluated with a questionnaire at postintervention regarding participants' satisfaction with applying and wearing the accelerometers during the intervention
Improvement of physical activity | 8 weeks
  Evaluation of improvement of habitual physical activity, all participants wore axivity (AX3) (Axivity, Newcastle, UK) accelerometers for seven consecutive days before, during and after the intervention. Accelerometer data was considered valid if the participant had minimum 22 hours wear time out of 24 possible. A measurement period was considered valid, if the participant had at least three valid weekdays and one valid weekend day. Any improvement in habitual physical activity (daily counts per minute) from baseline to postintervention was considered as an improvement
Adverse events | 8 weeks
  Evaluation of adverse events involved experienced severity of adverse events in the postintervention questionnaire according to the Patient-Reported Outcomes version of the Common Terminology Criteria for Adverse Events (PRO-CTCAE®).
  Minor adverse events covered dizziness, acute and prolonged musculoskeletal pain, and minor falls. Serious adverse events covered life-threatening events, disability, permanent damage, or hospitalization

SECONDARY OUTCOMES:
Questionnaires | 8 weeks
  1. Change in behavioral physical activity measured using a weekly questionnaire and compared at baseline and post-intervention
  2. Change in mental well-being measured using a weekly questionnaire and compared at baseline and post-intervention. Self-reported mental well-being were obtained with the World Health Organization( WHO)-5-Well-Being-Index Health-Related Quality of Life ( HRQoL). Questions were scored from 0 (none of the time) to 5 (all time).
     According to the recommendations, the raw score is multiplied by 4 to obtain a percentage score ranging from 0-100. The score was interpreted as following: 2.1. A score <50 was categorized as low HRQoL and described as being at risk for developing stress and depression 2.2. A score ≥50 was categorized as moderate to high HRQoL
  3. Change in physical activity measured using a weekly questionnaire and compared at baseline and post-intervention

CONTACTS AND LOCATIONS:
Overall Officials: Mathias R Larsen, PhD, Principal Investigator — Center for Physical Activity Research, Copenhagen University Hospita
Locations (1):
- Center for Physical Activity Research, Copenhagen, København N, Denmark

IPD SHARING:
Plan to Share IPD: Undecided
If the data can be fully anonymized the data can be shared

REFERENCES:
- [Derived] Mortensen SR, Pedersen ME, Skou ST, Ried-Larsen M. Online Physical Exercise and Group Sessions to Increase and Maintain Physical Activity in Individuals with Type 2 Diabetes: A Single-Arm Feasibility Study. Int J Environ Res Public Health. 2023 Feb 7;20(4):2893. doi: 10.3390/ijerph20042893. PMID 36833589